CLINICAL TRIAL: NCT00344383
Title: An Open-Label Study Evaluating the Bleeding Profile of Ortho Tri-Cyclen Lo (Norgestimate/Ethinyl Estradiol) Administered as an Extended Regimen
Brief Title: An Open-Label Study Evaluating Breakthrough Bleeding and Spotting With Norgestimate/Ethinyl Estradiol Tablets Administered as an Extended Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR008344
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Metrorrhagia
Keywords: oral contraceptive; breakthrough bleeding; spotting
MeSH Terms: conditions — Metrorrhagia | interventions — Moxifloxacin

INTERVENTIONS:
Drug: Norgestimate/Ethinyl Estradiol tablet

SUMMARY:
The purpose of this study is to evaluate the bleeding profile of norgestimate/ethinyl estradiol, an oral contraceptive tablet, given in an extended regimen

DETAILED DESCRIPTION:
This is an open-label study evaluating the bleeding profile of norgestimate/ethinyl estradiol tablets administered as an extended regimen (84 consecutive days of active tablets followed by seven days medication free) following a traditional regimen of two 28-day cycles (21 days of active tablets, followed by seven days of placebo tablets) of norgestimate/ethinyl estradiol tablets. All patients will receive norgestimate/ethinyl estradiol tablets in a traditional regimen for two 28-day cycles. Following the Traditional Treatment Phase, all patients will receive norgestimate/ethinyl estradiol tablets in an Extended Regimen Treatment Phase, consisting of 84 days of treatment with norgestimate/ethinyl estradiol tablets. Safety evaluations include physical examinations, adverse event reporting and vital signs. The hypothesis of the study is that a triphasic extended regimen would not result in breakthrough bleeding and spotting when the progestin dose drops. Traditional Regimen: two 28 day cycles of norgestimate 180 mcg daily for 1 week, 215 mcg daily for 1 week, 250 mcg daily for 1 week, placebo daily for 1 week. Extended Regimen: four uninterrupted cycles of norgestimate 180 mcg daily for 1 week, 215 mcg daily for 1 week, 250 mcg daily for 1 week, 1 week medication-free. In both Treatment Regimens patients receive ethinyl estradiol 25 mcg in each active tablet. The study is 147 days, Traditional days 1-56 and Extended days 57-147

ELIGIBILITY:
Inclusion Criteria:

* Subjects in good health as confirmed by medical history, physical exam, and PAP smear within the preceding six months
* Non-smokers, if between 35 and 45 years of age
* Patients who are not pregnant or lactating
* Had at least one normal menstrual period within 35 days prior to screening
* Completed their last term pregnancy at least 42 days prior to screening and had at least one normal menstrual period since the last pregnancy
* Must be post-menarcheal (have had at least one normal menstrual period) and pre-menopausal (having regular menstrual periods)

Exclusion Criteria:

* History or presence of disorders commonly accepted as contraindications to steroid hormonal therapy, eg, menopause, active or history of deep vein thrombophlebitis, thromboembolic disorders or hypercoagulation disorders, cerebral vascular or coronary artery disease, uncontrolled hypertension, or migraines with focal aura, benign or malignant liver tumor that developed during the use of oral contraceptives or estrogen-containing products
* carcinoma of any body system, diabetes mellitus with vascular involvement, known or suspected estrogen-dependent neoplasia, cholestatic jaundice, undiagnosed abnormal vaginal bleeding, neurovascular lesion of the eye, clinically relevant impairment of liver function, liver disease or renal disease
* absence of cyclic bleeding for at least three months, recent history of alcohol or other substance abuse
* significant depression or psychiatric disease that would result in an unreliable patients
* any subject deemed by the investigator to have questionable reliability in her ability to comply with the protocol and provide accurate information.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2003-11; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variables include the number of breakthrough bleeding and/or spotting days during the extended regimen treatment phase and the number of breakthrough bleeding days during the extended regimen treatment phase.

SECONDARY OUTCOMES:
Secondary efficacy variables include the number of bleeding and/or spotting days, number of bleeding days, number of bleeding and/or spotting episodes, and number of bleeding episodes during both treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.